CLINICAL TRIAL: NCT05038501
Title: Prevalence of Comorbidities in Patients Undergoing Oncosurgeries at Tertiary Cancer Institute in North India
Acronym: oncosurgery
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Senior Consultant, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RGCI \ MK 1967
Record Dates: First submitted 2021-08-15; First posted 2021-09-09 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Comorbidities and Coexisting Conditions
Keywords: comorbidities; oncosurgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comorbidities in Oncosurgery patients: Prevalence of comorbidities as Coronary artery disease, Hypertension , Diabetes Mellitus,Hypothyroidism and Corona Virus Infection will be studied in patients undergoing Oncosurgeries.
  Interventions: Other: To study comorbidities in patients undergoing Oncosurgeries

INTERVENTIONS:
Other: To study comorbidities in patients undergoing Oncosurgeries — In the Preoperative Anaesthesia checkup we will study prevalence of comorbidities as Coronary artery Disease, Hypertension, Diabetes Mellitus , Hypothyroidism and prior Corona Virus Infection in patients undergoing Oncosurgeries

SUMMARY:
Investigators plan to study the prevalence of comorbidities in patients undergoing oncosurgeries

DETAILED DESCRIPTION:
Plan to study the prevalence of Coronary Artery Disease, Hypertension, Diabetes Mellitus, Hypothyroidism, History of Corona Virus infection in patients undergoing oncosurgeries.

In the Pre anesthesia checkup patients age , sex , Weight in kilograms, Height in centimeters , pulse rate, Blood Pressure will be noted and value>140/90 mmHg will be taken as hypertensive. History will be obtained about diagnosed Coronary Artery Disease , Diabetes Mellitus, Hypertension , Hypothyroidism , History of previous Corona Virus Infection (RT-PCR Test Positive) .Relevant investigations Electrocardiography and Echocardiography for assessment of Coronary Artery Disease. Fasting or Random Blood Sugar , Thyroid Function Test will be done .

Fasting Blood Sugar >126 milligram/ Decilitre and Random Blood sugar >200mg/dL will be taken as diabetic. TSH more than 5 micro IU/mL will be hypothyroid .

ELIGIBILITY:
Inclusion Criteria: Patients undergoing Oncosurgeries Age above 40 years .

-

Exclusion Criteria:

Age below 40 years Emergency Surgery Patient Refusal

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing Oncosurgeries will be studied for prevalence of comorbidites.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
To study Coronary Artery disease in patients undergoing Oncosurgeries | 60 days
  Electrocardiography and Echocardiography will be performed.
  Investigators will measure Blood Pressure , Blood Sugar , Thyroid Function Test and previous Corona Virus Infection
To study Diabetes Mellitus in patients undergoing Oncosurgeries. | 60days
  Random Blood Sugar in milligram/Decilitre will be measured.

SECONDARY OUTCOMES:
To study Hypothyroidism in patients undergoing Oncosurgeries | 60 days
  Thyroid Stimulating Hormone (TSH) in micro IU / millilitre will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kulkarni, MD, Principal Investigator — Rajiv Gandhi Cancer Institute and RC , Delhi, INDIA
Locations (1):
- Anita Kulkarni, Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta R, Mohan I, Narula J. Trends in Coronary Heart Disease Epidemiology in India. Ann Glob Health. 2016 Mar-Apr;82(2):307-15. doi: 10.1016/j.aogh.2016.04.002. PMID 27372534
- [Background] Ranasinghe P, Jayawardena R, Gamage N, Sivanandam N, Misra A. Prevalence and trends of the diabetes epidemic in urban and rural India: A pooled systematic review and meta-analysis of 1.7 million adults. Ann Epidemiol. 2021 Jun;58:128-148. doi: 10.1016/j.annepidem.2021.02.016. Epub 2021 Mar 13. PMID 33727086